CLINICAL TRIAL: NCT06599801
Title: The Clinical Outcomes of Thoracodorsal Artery Flap in Oral and Maxillofacial Defect Reconstruction: a Retrospective Study
Brief Title: Clinical Outcomes of Thoracodorsal Artery Flap in Oral and Maxillofacial Reconstruction
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-710-01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC)
Keywords: Oral Squamous Cell Carcinoma; thoracodorsal artery perforator flap; quality of life; free flap
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Anterolateral thigh flap group: Oral squamous cell carcinoma patients received the reconstruction with anterolateral thigh flaps after tumor resection
  Interventions: Procedure: Anterolateral thigh flap reconstruction surgery
- Forearm flap group: Oral squamous cell carcinoma patients received the reconstruction with forearm flaps after tumor resection
  Interventions: Procedure: Forearm flap reconstruction surgery
- Latissimus dorsi flap group: Oral squamous cell carcinoma patients received the reconstruction with latissimus dorsi flaps after tumor resection
  Interventions: Procedure: Forearm flaps reconstruction surgery
- Fibula flap group: Oral squamous cell carcinoma patients received the reconstruction with Fibula flaps after tumor resection
  Interventions: Procedure: Fibula flap reconstruction surgery
- Thoracodorsal artery perforator flap group: Oral squamous cell carcinoma patients received the reconstruction with Thoracodorsal artery perforator flaps after tumor resection
  Interventions: Procedure: Thoracodorsal artery perforator flap reconstruction surgery

INTERVENTIONS:
Procedure: Thoracodorsal artery perforator flap reconstruction surgery — Oral squamous cell carcinoma patients underwent reconstruction with thoracodorsal artery perforator (TDAP) flaps following tumor resection.
  Groups: Thoracodorsal artery perforator flap group
Procedure: Forearm flaps reconstruction surgery — Oral squamous cell carcinoma patients received the reconstruction with forearm flaps after tumor resection
  Groups: Latissimus dorsi flap group
Procedure: Anterolateral thigh flap reconstruction surgery — Oral squamous cell carcinoma patients received the reconstruction with anterolateral thigh flaps after tumor resection
  Groups: Anterolateral thigh flap group
Procedure: Fibula flap reconstruction surgery — Oral squamous cell carcinoma patients received the reconstruction with fibula flaps after tumor resection
  Groups: Fibula flap group
Procedure: Forearm flap reconstruction surgery — Oral squamous cell carcinoma patients received the reconstruction with forearm flaps after tumor resection
  Groups: Forearm flap group

SUMMARY:
The goal of this study is to retrospectively compare different types of free flaps to determine the most suitable free flap for functional reconstruction in oral squamous cell carcinoma patients following tumor resection. The main questions it aims to answer are:

Do the clinical characteristics of the thoracodorsal artery perforator flap differ from those of other types of flaps? Does the thoracodorsal artery perforator flap result in better clinical outcomes compared to other types of flaps? After reconstruction with the thoracodorsal artery perforator flap, do patients have better quality of life, speech function and scar healing compared to other types of flaps? Investigators will retrospectively compare the thoracodorsal artery perforator flap with other types of flaps (such as the anterolateral thigh flap, forearm flap, latissimus dorsi flap and fibula flap) to explore the most suitable free flap for facial defect reconstruction in oral squamous cell carcinoma patients.

Participants are oral squamous cell carcinoma patients who previously underwent facial defect reconstruction with different types of flaps. Participants have completed relevant questionnaires at 1, 3, 6 and 12 months post-surgery. The data will be scored and assessed by the investigators.

DETAILED DESCRIPTION:
Oral squamous cell carcinoma (OSCC) severely impacts patients's quality of life (QoL). The combined treatment approach of surgery, radiation and chemotherapy can lead to oral function impairments, including swallowing and speech difficulties. Postoperatively, patients may also experience physical, emotional and functional sequelae, resulting in a significant decline in their QoL.

Functional maxillofacial defect repair has become a mainstream approach in surgical reconstruction. The thoracodorsal artery perforator (TDAP) flap is increasingly favored by oral and maxillofacial surgeons due to its advantages of fewer complications, favorable tissue characteristics and easy access to the latissimus dorsi nerve, making it the preferred option for maxillofacial defect reconstruction.

Postoperative QoL has become an important indicator for evaluating the prognosis of OSCC. In successful cases of OSCC surgery, patients may still experience a decline in QoL due to postoperative complications, oral function impairments and aesthetic issues, leading to a suicide rate much higher than that of other cancer patients. Compared to traditional free flaps, the TDAP flap has less conspicuous donor site scarring, which is hidden under the posterior axillary fold, thus offering significant advantages in aesthetics. Additionally, the motor nerve of the TDAP flap helps achieve functional reconstruction of the maxillofacial area, improving the postoperative QoL for OSCC patients.

In this retrospective study, the investigators will collect clinical data from 217 OSCC patients who underwent different free flap reconstructions at the Oral and Maxillofacial Surgery Department of Sun Yat-sen Memorial Hospital from January 2020 to December 2023. The investigators will assess the QoL, speech ability and scarring of patients using the Washington Quality of Life Scale, Speech Disorder Index Scale and Vancouver Scar Scale. The goal is to evaluate the repair and reconstruction outcomes of the TDAP flap in OSCC patients and to identify the most suitable flap choice for OSCC patients at this stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with oral squamous cell carcinoma who have completed comprehensive imaging examinations before surgery.
2. Preoperative pathological biopsy confirmed as oral squamous cell carcinoma.
3. Patients with oral squamous cell carcinoma who have completed comprehensive laboratory tests before surgery.
4. Patients with oral squamous cell carcinoma who underwent tumor resection and flap reconstruction at our hospital.
5. Postoperative pathological diagnosis confirmed as oral squamous cell carcinoma.
6. Patients with oral squamous cell carcinoma who attend follow-up visits at 1, 3, 6, and 12 months post-surgery, completing all clinical examinations and questionnaires.

Exclusion Criteria:

1. Patients with oral squamous cell carcinoma who lack imaging data or have artifacts affecting imaging results.
2. Patients with oral squamous cell carcinoma who have incomplete laboratory test results from our hospital.
3. Patients with oral squamous cell carcinoma with postoperative pathology that remains unclear or cannot be confirmed as oral squamous cell carcinoma.
4. Patients with oral squamous cell carcinoma who are unable to attend follow-up visits at 1, 3, 6, and 12 months.
5. Patients who do not complete the questionnaires as required during follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with oral squamous cell carcinoma undergoing reconstruction with thoracodorsal artery perforator flap, anterolateral thigh flap, forearm flap, latissimus dorsi flap, or fibula flap at Sun Yat-sen Memorial Hospital of Sun Yat-sen University from January 2020 to June 2023 will be included. Descriptive statistics will be generated for all outcome measures. Statistical analysis will be conducted using SPSS software version 23.0.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Quality of Life | Postoperative at 1, 3, 6, and 12 months
  The investigators applied the University of Washington Quality of Life (UW-QOL) questionnaire to evaluate the participants' appearance, functional outcomes and emotional well-being. This included scores for pain, appearance, activity, comfort, swallowing, chewing, speech, shoulder function, taste, saliva, emotion, anxiety and the overall total score. According to the UW-QOL version 4 questionnaire, each domain is scored on a scale from 0 to 100, with higher scores indicating a better quality of life.
Postoperative Speech Function | Postoperative at 1, 3, 6, and 12 months
  The investigators evaluated postoperative speech function using the 30-item Speech Handicap Index (SPI) questionnaire. This questionnaire employs a 5-point Likert scale with the following response categories: "never" (0 points), "almost never" (1 point), "sometimes" (2 points), "almost always" (3 points), and "always" (4 points). The total SPI score ranges from 0 to 120 and includes two subscales: psychosocial function and speech function, each consisting of 14 items. Lower scores indicate better speech function.
Scar Assessment | Postoperative at 1, 3, 6, and 12 months
  The investigators applied the Vancouver Scar Scale (VSS) questionnaire to evaluate the participants' scars at the donor site. This included scores for the pigmentation (score from 0-3), thickness (score from 0-3), blood supply (score from 0-5) and texture (score from 0-3) of the scar at donor site. According to the VSS questionnaire, a lower score indicates a better outcome with the similar appearance like normal, however a higher score indicates an abnormal appearance and contracture.
Swallowing Function Assessment | Postoperative at 1, 3, 6, and 12 months
  The investigators applied the NIH Swallowing Safety Scale (NIH-SSS) questionnaire to evaluate the participants' swallowing function. The total score of NIH-SSS ranges from 0 to 10 points, with each score reflecting a different level of swallowing safety. A score of 0 indicates completely safe swallowing with no signs of aspiration or difficulty, while a score of 10 represents the most severe aspiration or swallowing impairment, potentially requiring urgent intervention.

SECONDARY OUTCOMES:
Flap Complication Incidence | Postoperative at 1, 3, 6, and 12 months
  The rate at which the blood supply to the flap suddenly interrupts or significantly decreases postoperatively, leading to ischemia or necrosis of the flap.
Flap Failure Incidence | Postoperative at 1, 3, 6, and 12 months
  The rate at which the flap fails to survive and heal due to insufficient blood supply, infection, technical issues, or other complications, resulting in partial or complete necrosis of the flap.
Postoperative Complications | Postoperative at 1, 3, 6, and 12 months
  Includes complications at the recipient site (hematoma, infection, wound dehiscence, and fistula), complications at the donor site (hematoma, infection, and wound dehiscence), and lower limb venous thrombosis.
Patient Bed Rest Duration | Postoperative at 1 months
  The time a patient spends completely resting in bed postoperatively, during which the patient is unable to move independently or can only perform necessary bedside activities with the assistance of caregivers.
Flap Pedicle Vein Diameter | Postoperative at 1 day
  The investigators used a Micro-Vessel Caliper to measure the cross-sectional diameter of the vein in the flap pedicle during flap-harvesting surgery.
Flap Pedicle Artery Diameter | Postoperative at 1 day
  The investigators used a Micro-Vessel Caliper to measure the cross-sectional diameter of the artery in the flap pedicle during flap-harvesting surgery.
Flap Pedicle Vessel Separation Length | Postoperative at 1 day
  The maximum distance that can be separated between the point where the flap's blood supply vessel (artery or vein) enters the flap and the furthest point of its branching.
Flap Surgical Operation Time | Postoperative at 1 day
  The total time spent on the flap procedure, including the time for designing the flap, harvesting the flap, shaping the flap, and placing and securing the flap.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen Univerity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
To protect participants' privacy, the data may include sensitive information such as personal identification or health status. If IPD is needed, please contact the project investigator.

REFERENCES:
- [Background] Min F, Qiu P, Zhu X, Zhou B, Lin Z, Pan C, Wang Y. Modified submandibular mandibulotomy approach versus lip-splitting approach in tongue cancer surgery: a retrospective paired-cohort study. Clin Oral Investig. 2023 Dec 26;28(1):32. doi: 10.1007/s00784-023-05395-3. PMID 38147089
- [Background] Zhou B, Liao J, Zhu C, Yuan K, Liu Z, Lin Z, Huang Z, Chen W, Li J, Wang Y. Full cheek defect reconstruction using ALTF versus RFF: Comparison of quality of life, clinical results, and donor site morbidity. Oral Dis. 2020 Sep;26(6):1157-1164. doi: 10.1111/odi.13354. Epub 2020 May 4. PMID 32289869
- [Derived] Wu F, Xia X, Zhu C, Fu M, Zhu X, Wang J, Lan T, Wang Y. Functional tongue reconstruction using innervated TDAP versus ALT free flaps: a retrospective paired-cohort study. Head Face Med. 2025 Dec 5;22(1):3. doi: 10.1186/s13005-025-00572-z. PMID 41350686